CLINICAL TRIAL: NCT06452628
Title: Effects of Mulligan Mobilizations Versus Active Release Technique on Pain, Range of Motion and Disability in Patients With Tension-Type Headache.
Brief Title: Mulligan Mobilizations Versus Active Release Technique in Tension-type Headache.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ RCR & AHS/23/01107
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Mulligan Mobilizations; Active release technique; cervical spine; manual therapy
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial.
Who Masked: Outcomes Assessor
Masking Description: Blinding refers to a practice where study participants are prevented from knowing certain information that may somehow influence them-thereby tainting the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): This group will receive Mulligan mobilizations.
  Interventions: Other: Mulligan mobilizations
- Group B (Active Comparator): This group will receive the Active release technique.
  Interventions: Other: Active Release Technique
- Group C (Other): This group will receive both techniques combined.
  Interventions: Other: Mulligan mobilizations with active release technique

INTERVENTIONS:
Other: Mulligan mobilizations — The duration of the intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with Mulligan mobilizations.
  Arms: Group A
Other: Active Release Technique — The duration of the intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with the Active release technique.
  Arms: Group B
Other: Mulligan mobilizations with active release technique — The duration of intervention will be 4 weeks, 3 sessions a week, a total of 12 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with mulligan mobilizations with active release technique.
  Arms: Group C

SUMMARY:
Tension-type headaches, characterized by a dull, aching head pain, are one of the most prevalent forms of headache disorders worldwide. Although they are typically not associated with severe disability or neurological symptoms, they can significantly impact an individual's quality of life due to chronic pain and discomfort. Non-pharmacological interventions, such as manual therapy techniques, have gained prominence in headache management, offering potential relief and functional improvements for patients. This study aims to investigate the comparative effectiveness of two widely used manual therapy approaches, Mulligan mobilization and Active Release Technique (ART), in alleviating pain, reducing disability, and enhancing range of motion (ROM) in patients suffering from tension-type headaches. Understanding which technique offers superior outcomes is vital for optimizing headache management strategies.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will recruit adult participants diagnosed with tension-type headaches according to standardized criteria. Eligible individuals will be randomly assigned to one of three groups: The Mulligan mobilization group, the ART group, and the control group. Each group will undergo a specific manual therapy intervention protocol administered by trained therapists. The primary outcome measures will include assessments of pain intensity via VAS, disability levels via Headache disability index (HDI), Stress levels will be assessed by PSS (Perceived Stress Scale), and ROM of the cervical spine by using the Flexion rotation test. Secondary outcomes will encompass patient-reported measures of headache frequency, medication usage, and overall quality of life. Data will be collected at baseline, immediately post-intervention, and at follow-up intervals. Statistical analyses will be conducted to assess and compare the effects of the two interventions on the primary and secondary outcomes using ANOVA from SPSS software, thereby addressing the research question regarding their relative efficacy. This study holds the potential to enhance the evidence base for non-pharmacological headache management and guide clinicians and patients toward more effective treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-35 years.
* Diagnosis of chronic tension-type headache according to the International Classification of --Headache Disorders (ICHD-3) criteria.
* Baseline HDI from 10 and above, and NPRS score 3 and above.
* No prior exposure to any of the two interventions (ART and Mulligan Mobilization).

Exclusion Criteria:

* All other types of headaches.

  * Individuals taking medications for headaches.
  * Serious neurological or medical conditions that could affect the study outcomes.
  * History of psychiatric disorders.
  * Recent head or neck trauma or surgery.
  * Contraindications for any of the two interventions.
  * Participation in other headache management studies during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain: Numeric Pain Rating Scale(NPRS) | 4th week
  Changes from baseline Numeric pain rating scale is The 11-point scale used to capture the patient's level of pain. The scale is anchored on the left with the phrase ''no pain'' and on the right with the phrase ''worst imaginable pain.'' Patients rate their current level of pain and their worst and least amount of pain in the last 24 hours. Numeric pain scales have been shown to be reliable and valid with validity range from 0.86 to 0.95 and high test-retest reliability r=0.96.
Disability: Headache Disability Index(HDI) | 4th week
  Changes from baseline the Headache Disability Index (HDI) is a valid and reliable questionnaire designed to assess the impact of headaches on daily functioning and activities. It is often used to quantify the level of disability associated with headaches. The HDI consists of 25 items, and each item is scored on a scale from 0 to 6.
Range of motion Cervical(Flexion) | 4th week
  Changes from the baseline ROM range of motion of cervical flexion will be taken with the help of a universal goniometer.
Range of motion Cervical(Extension) | 4th week
  Changes from the baseline ROM range of motion of cervical extension will be taken with the help of universal goniometer.
Range of motion Cervical(Rotation) | 4th week
  Changes from the baseline ROM range of motion of cervical rotation will be taken with the help of a universal goniometer.
Range of motion Cervical(Side bending) | 4th week
  Changes from the baseline ROM range of motion of cervical side bending will be taken with the help of a universal goniometer.

OTHER OUTCOMES:
Stress: Perceived Stress Scale(PSS) | 1st week
  Changes from the baseline the Perceived Stress Scale (PSS) is a classic stress assessment instrument. The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certain way For each question choose from the following alternatives: 0 - never, 1 - almost never, 2 - sometimes, 3 - fairly often, 4 - very often

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hajra, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital Toba Tek Singh, Toba Tek Singh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashina S, Mitsikostas DD, Lee MJ, Yamani N, Wang SJ, Messina R, Ashina H, Buse DC, Pozo-Rosich P, Jensen RH, Diener HC, Lipton RB. Tension-type headache. Nat Rev Dis Primers. 2021 Mar 25;7(1):24. doi: 10.1038/s41572-021-00257-2. PMID 33767185
- [Background] Jensen RH. Tension-Type Headache - The Normal and Most Prevalent Headache. Headache. 2018 Feb;58(2):339-345. doi: 10.1111/head.13067. Epub 2017 Mar 13. PMID 28295304
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Fernandez-de-Las-Penas C, Florencio LL, Plaza-Manzano G, Arias-Buria JL. Clinical Reasoning Behind Non-Pharmacological Interventions for the Management of Headaches: A Narrative Literature Review. Int J Environ Res Public Health. 2020 Jun 9;17(11):4126. doi: 10.3390/ijerph17114126. PMID 32527071
- [Background] Burch R. Migraine and Tension-Type Headache: Diagnosis and Treatment. Med Clin North Am. 2019 Mar;103(2):215-233. doi: 10.1016/j.mcna.2018.10.003. Epub 2018 Dec 3. PMID 30704678
- [Background] Robbins MS. Diagnosis and Management of Headache: A Review. JAMA. 2021 May 11;325(18):1874-1885. doi: 10.1001/jama.2021.1640. PMID 33974014
- [Background] Del Blanco Muniz JA, Zaballos Laso A. [Tension-type headache. Narrative review of physiotherapy treatment]. An Sist Sanit Navar. 2018 Dec 26;41(3):371-380. doi: 10.23938/ASSN.0379. Spanish. PMID 30425380
- [Background] McDowell JM, Johnson GM, Hetherington BH. Mulligan Concept manual therapy: standardizing annotation. Man Ther. 2014 Oct;19(5):499-503. doi: 10.1016/j.math.2013.12.006. Epub 2014 Jan 10. PMID 24491791